CLINICAL TRIAL: NCT00104117
Title: A Phase 1 Dose Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL999 Administered Intravenously to Subjects With Solid Tumors
Brief Title: Study of XL999 in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-001
Record Dates: First submitted 2005-02-23; First posted 2005-02-24 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — XL999 was to be given biweekly to an initial cohort of subjects at 0.20 mg/kg and to successive cohorts at doses that escalated by cohort according to a design for safely determining an MTD. After determination of the MTD, one or more additional cohorts were to receive XL999 weekly at the MTD or a lower dose, as determined by the CRC on the basis of interim safety and PK data. By a protocol amendment after initiation of the study, subjects were to be enrolled in an additional cohort to receive a weekly XL999 dose of 200 mg.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of XL999 in adults with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Cancer that has progressed on currently available therapies
* Life expectancy of >3 months
* Adequate bone marrow, liver, and kidney function
* Willing to use accepted method of contraception during the course of the study
* Negative pregnancy test (females)
* Written informed consent

Exclusion Criteria:

* Chemotherapy within 4-6 weeks of the start of treatment (depending on the therapy)
* Radiotherapy within 4 weeks of the start of treatment
* Subjects with known brain metastasis
* Uncontrolled medical disorder such as infection or cardiovascular disease
* Subjects known to be HIV positive
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-11; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and to assess the safety and tolerability of XL999 administered as a single 4-hour intravenous (IV) infusion in subjects with solid tumors | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
To evaluate plasma pharmacokinetics (PK) and estimate renal elimination of XL999 administered as a single 4-hour IV infusion in subjects with solid tumors | Various timepoints from pre-dosing until 48 hours post dose.
To evaluate the PK of XL999 administered at a fixed weekly dose of 200 mg. | At various timepoints from pre-dosing until 48 hours post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Paul Woodard, MD, Study Director — Exelixis
Locations (2):
- United States (2):
  - Case Western Reserve University, Univserzity Hospitals of Cleveland, Cleveland, Ohio
  - Cancer Therapy and Research Center, Institute for Drug Development, San Antonio, Texas